CLINICAL TRIAL: NCT05165381
Title: Video Plethysmography for Contactless Vital Signs Measurement: A Pilot Study
Brief Title: Contactless Vital Signs Measurement
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 21-6075
Record Dates: First submitted 2021-12-10; First posted 2021-12-21 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Blood Pressure, Heart Rate, Respiratory Rate, Heart Rate Variability, Stress Index, Vital Signs Monitoring; Vital Signs Monitoring
Keywords: vital signs

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Contactless vital signs and stress measurement.: Contactless vital signs and stress measurement. Eligible participants will agree to have a 1.5-minute facial video recorded using an iPad. Video will be processed through a specialized algorithm to obtain BP, HR, RR, HRV and stress index. measurements.
  Interventions: Device: Video PPG

INTERVENTIONS:
Device: Video PPG — Contactless vital signs and stress measurement using video PPG technology. An iPad will be used to record a video of the participant's, which can then be converted to vital signs using a specialized algorithm.

SUMMARY:
This pilot study will determine the feasibility and effectiveness of implementing video plethysmography (PPG) for contactless vital signs and str5ess index measurements from surgical patients in preoperative care. Our primary objective is to determine the feasibility and validity of using video PPG to collect contactless BP, HR and RR measurements when compared medical-grade instruments. Our secondary objective is to validate the use of video PPG in measuring HRV and stress index when compared to a validated stress questionnaire.

DETAILED DESCRIPTION:
The huge impact of the COVID-19 pandemic on global healthcare systems has given rise to an increased need for virtual care. This pilot study will determine the feasibility and effectiveness of implementing video plethysmography (PPG)for contactless vital signs measurements such as blood pressure (BP), heartrate (HR), respiratory rate (RR) and heart rate variability (HRV) from surgical patients in preoperative care. We also aim to validate the use of video PPG in measuring HRV and stress index when compared to a validated stress questionnaire.

This study aims to assess how video PPG technology can be implemented in a clinical and telemedicine. If proven to be effective, this technology can be integrated into any smartphone or tablet and will allow users to monitor their vital signs with just a 1.5-minute video.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective ambulatory surgery with general and/or regional anesthesia;
* 18 years or older;
* able to comprehend study instructions in English

Exclusion Criteria:

* refusal to consent for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergoing elective inpatient surgery under general and/or regional anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Vital signs measurement | 24 hours
  Blood pressure will be measured by using both video PPG and standard medical grade blood pressure machine preoperatively
Vital signs measurement | 24 hours
  Heart rate will be measured by using both video PPG and standard medical grade blood pressure machine preoperatively.[
Vital signs measurement | 24 hours
  Breathing rate will be measured by using both video PPG and standard medical grade blood pressure machine preoperatively
HRV and stress index pressure | 24 hours
  4. HRV and stress index pressure will be measured by video PPG, stress index will be measured with a validated questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Frances Chung, MBBS FRCPC, Principal Investigator — University Health Network, Toronto Western Hospital
Locations (2):
- Canada (2):
  - 399 Bathurst St.,Toronto Western Hopsital, Preadmission Clinic, Dept. of Anesthesia, Toronto, Ontario
  - University Health Network, Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pham C, Poorzargar K, Panesar D, Lee K, Wong J, Parotto M, Chung F. Video plethysmography for contactless blood pressure and heart rate measurement in perioperative care. J Clin Monit Comput. 2024 Feb;38(1):121-130. doi: 10.1007/s10877-023-01074-6. Epub 2023 Sep 16. PMID 37715858